CLINICAL TRIAL: NCT00554229
Title: A Phase III Trial to Test the Efficacy of ZD4054(Zibotentan), an Endothelin A Receptor Antagonist, Versus Placebo in Patients With Hormone Resistant Prostate Cancer (HRPC) and Bone Metastasis Who Are Pain Free and Mildly Symptomatic.
Brief Title: A Phase III Trial of ZD4054 (Zibotentan) (Endothelin A Antagonist) in Hormone Resistant Prostate Cancer With Bone Metastases
Acronym: ENTHUSE M1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4320C00014; 2007-003227-20 (EudraCT Number); NCT00707395 (obsolete NCT alias)
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: Hormone Resistant Prostate Cancer; Endothelin A Receptor Antagonist; Endothelin A; Endothelin A antagonist
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZD4054 (Experimental): ZD4054 10 mg oral tablet once daily
  Interventions: Drug: ZD4054
- Placebo (Placebo Comparator): Matching Placebo, oral tablets once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZD4054 — ZD4054 10 mg oral tablet once daily
  Other Names: Zibotentan
  Arms: ZD4054
Drug: Placebo — Matching placebo oral tablet once daily
  Arms: Placebo

SUMMARY:
Enthuse M1 is a large phase III clinical trial studying the safety and efficacy of ZD4054 (Zibotentan) in patients with hormone resistant prostate cancer and bone metastases.

* This clinical trial will test if the Endothelin A Receptor Antagonist ZD4054 (Zibotentan) can improve survival compared with placebo.
* ZD4054(Zibotentan) is a new type of agent, which is thought to slow tumour growth and spread by blocking Endothelin A receptor activity. This trial will look at the effects of ZD4054 (Zibotentan) in hormone resistant prostate cancer patients with bone metastases.
* All patients participating in this clinical trial will receive existing standard prostate cancer treatments in addition to trial therapy.
* Half the patients will receive ZD4054 (Zibotentan), and half the patients will receive placebo in addition to standard prostate cancer therapy. By participating in this trial there is a 50% chance that patients will receive an agent that may slow the progression of the tumour.
* No patients will be deprived of standard prostate cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients who answer TRUE to the following criteria may be eligible to participate in this trial.

1. Confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate) that has spread to the bone (bone metastases)
2. Increasing Prostate Specific Antigen (PSA) over a one month period
3. No pain, or mild pain from prostate cancer
4. Currently receiving treatment with surgical or medical castration

Exclusion Criteria:

Patients who answer TRUE to the following may NOT eligible to participate in this trial.

1. Currently using opiates based pain killers)
2. Previous treatment with chemotherapy (paclitaxel, docetaxel, and mitoxantrone)
3. Suffering from heart failure or had a myocardial infarction within last 6 months
4. A history of epilepsy or seizures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gleave, MD, FRCSC, FACS, Principal Investigator — The Prostate Centre at Vancouver General Hospital; Joel B Nelson, MD, Principal Investigator — University of Pittsburgh
Locations (197):
- United States (19):
  - Research Site, Tucson, Arizona
  - Research Site, Greenbrae, California
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California
  - Research Site, San Mateo, California
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainsville, Florida
  - Research Site, Port St.Lucie, Florida
  - Research Site, Des Moines, Iowa
  - Research Site, Canton, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Wheeling, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (2):
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Santa Fe, Santa Fe Province
- Australia (5):
  - Research Site, Hornsby, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Redcliffe, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Subiaco, Western Australia
- Austria (2):
  - Research Site, Graz, Graz
  - Research Site, Wels, Wels
- Belgium (4):
  - Research Site, Brussels, Brussels Capital
  - Research Site, Ghent, Gent
  - Research Site, Kortrijk, Kortrijk
  - Research Site, Leuven, Leuven
- Brazil (8):
  - Research Site, Fortaleza, Ceará
  - Research Site, Goiânia, Goiás
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Ribeirão Preto, São Paulo
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Canada (19):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Kentville, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Granby, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Point-Claire, Quebec
  - Research Site, Québec, Quebec
- China (9):
  - Research Site, Haidian District, Beijing Municipality
  - Research Site, XI Cheng District, Beijing Municipality
  - Research Site, Xicheng District, Beijing Municipality
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Pudong New Area, Shanghai Municipality
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xuhui District, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
- Czechia (4):
  - Research Site, Brno, Brno
  - Research Site, Olomouc, Olomouc
  - Research Site, Prague, Prague
  - Research Site, Ústí nad Labem, Usti nad Labem
- Denmark (4):
  - Research Site, Aalborg, Aalborg
  - Research Site, Aarhus, Aarhus
  - Research Site, Herlev, Herlev
  - Research Site, Copenhagen, Kobenhavn
- Finland (3):
  - Research Site, Joensuu, Joensuu
  - Research Site, Kajaanintie, Kajaanintie
  - Research Site, Tampere, Pirkanmaa
- France (6):
  - Research Site, Montpellier, Montpellier
  - Research Site, Paris, Paris
  - Research Site, Poitiers, Poitiers Cedex
  - Research Site, Suresnes, Suresnes
  - Research Site, Toulouse, Toulouse
  - Research Site, Villejuif, Villejuif
- Germany (11):
  - Research Site, Augsburg, Augsburg
  - Research Site, Bad Gegeberg, Bad Gegeberg
  - Research Site, Emmendingen, Emmendingen
  - Research Site, Leipzig, Leipzig
  - Research Site, Lübeck, Luebeck
  - Research Site, Mannheim, Mannheim
  - Research Site, München, Muenchen
  - Research Site, Planegg, Muenchen
  - Research Site, Reutlingen, Reutlingen
  - Research Site, Berlin, State of Berlin
  - Research Site, Kirchheim, Teck
- Hong Kong (3):
  - Research Site, Hong Kong, Hong Kong
  - Research Site, Tuenmen, Hong Kong
  - Research Site, Shatin, Shatin
- Hungary (5):
  - Research Site, Budapest, Budapest
  - Research Site, Debrecen, Debrecen
  - Research Site, Miskolc, Miskolc
  - Research Site, Nyíregyháza, Nyiregyhaza
  - Research Site, Szeged, Szeged
- India (11):
  - Research Site, Gujarat, Gujarat
  - Research Site, Trivandrum, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Rohini, National Capital Territory of Delhi
  - Research Site, New Delhi, New Delhi
  - Research Site, Chandigarh, Punjab
  - Research Site, Ludhiana, Punjab
  - Research Site, Bikaner, Rajasthan
  - Research Site, Jaipur, Rajasthan
  - Research Site, Kolkota, West Bengal
- Italy (2):
  - Research Site, Milan, Milan
  - Research Site, Rome, Rome
- Japan (28):
  - Research Site, Asahi, Chiba
  - Research Site, Chiba, Chiba
  - Research Site, Narashino, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Maebashi, Gunma
  - Research Site, Ōtake, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Kita-gun, Kagawa-ken
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Osaka, Osaka
  - Research Site, Ōsaka-sayama, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Wako, Saitama
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Fuchu_city, Tokyo
  - Research Site, Itabashi-Ku, Tokyo
  - Research Site, Meguro-ku, Tokyo
  - Research Site, Mitaka, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
- Mexico (3):
  - Research Site, Mexico City, Mexico City
  - Research Site, Distrito Federal Ciudad, Mexico
  - Research Site, Metepec, State of Mexico
- Netherlands (4):
  - Research Site, Amsterdam, Amsterdam
  - Research Site, Eindhoven, Eindhoven
  - Research Site, Nijmegen, Nijmegen
  - Research Site, Groningen, Provincie Groningen
- Poland (6):
  - Research Site, Bialystok, Bialystok
  - Research Site, Kościerzyna, Koscierzyna
  - Research Site, Krakow, Krakow
  - Research Site, Rzeszów, Rzeszow
  - Research Site, Warsaw, Warszawa
  - Research Site, Wroclaw, Wroclaw
- Portugal (3):
  - Research Site, Coimbra, Coimbra District
  - Research Site, Lisbon, Lisbon District
  - Research Site, Porto, Porto District
- Russia (8):
  - Research Site, Barnaul, Barnaul
  - Research Site, Stary Oskol, Belgorod Oblast
  - Research Site, Izhevsk, Izhevsk
  - Research Site, Kursk, Kursk Oblast
  - Research Site, Moscow, Moscow
  - Research Site, Saint Petersgurg, Saint Petersgurg
  - Research Site, Sochi, Sochi
  - Research Site, Voronezh, Voronezh Oblast
- Serbia (3):
  - Research Site, Belgrade, Belgrade
  - Research Site, Niš, Nis
  - Research Site, Novi Sad, Novi Sad
- Research Site, Singapore, Singapore, Singapore
- South Africa (4):
  - Research Site, Bloemfontein, Bloemfontein
  - Research Site, Tygerberg, Cape Town
  - Research Site, Pietermaritzburg, Pietermaritzburg
  - Research Site, Port Elizabeth, Port Elizabeth
- South Korea (5):
  - Research Site, Seo-gu, Busan
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Heungduk-gu Cheongju, North Chungcheong
  - Research Site, Gangnam-gu, Seoul
  - Research Site, Songpa-gu, Seoul
- Sweden (3):
  - Research Site, Gothenburg, Goteborg
  - Research Site, Gothenburg, Gothenburg
  - Research Site, Stockholm, Stockholm County
- Switzerland (4):
  - Research Site, Basel, Basel
  - Research Site, Bern, Canton of Bern
  - Research Site, Locarno, Locarno
  - Research Site, Sursee, Sursee
- Taiwan (3):
  - Research Site, Kaohsiung City, Kaohsiung
  - Research Site, Taipei, Taipei
  - Research Site, Taoyuan District, Taiwan
- United Kingdom (5):
  - Research Site, Reading, Berkshire
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, Maidstone, Kent
  - Research Site, London, London
  - Research Site, Huddersfield, Yorkshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 896 patients with hormone-resistant prostate cancer patients and bone metastasis were recruited between 20th November 2007 and 13th February 2009.
Pre-assignment Details: 302 of the 896 enrolled patients were not randomised to treatments groups as they failed screening.
Groups:
- Placebo: Placebo oral tablet once daily
Period: Overall Study
Arm/Group | ZD4054 | Placebo
Started | 299 | 295
Patients Who Received Treatment | 298 | 295
Completed | 73 | 70
Not Completed | 226 | 225
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 29 | 37
Not completed — Adverse Event | 71 | 39
Not completed — Protocol Violation | 3 | 3
Not completed — Reason not otherwise captured, eg; death | 119 | 140
Not completed — Randomised but no treatment received | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZD4054 | Placebo | Total
Number analyzed (Participants) | 299 | 295 | 594
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Overall | 70.2 (7.8) | 70.9 (8.6) | 70.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 299 | 295 | 594

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Median time (in months) from randomisation until death using the Kaplan-Meier method
Time Frame: From date of randomization until date of death, assessed up to 32 months
Measure: Median (Full Range); unit: months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
months | 24.5 [0.5 to 31.2] | 22.5 [0.5 to 29.8]

2. Secondary Outcome: Progression Free Survival
Description: Median time (in months) from randomisation until clinical progression of disease, where progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline, using the Kaplan-Meier method
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 31 months
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 6.2 [2.8 to 13.8] | 6.5 [2.8 to 13.2]

3. Secondary Outcome: Time to Use of Opiates
Description: Median time (in months) from randomisation until use of opiates for disease-related symptoms for a duration ≥1 week using the Kaplan-Meier method
Time Frame: From date of randomization until use of opiates for disease-related symptoms for a duration ≥1 week, assessed up to 31 months
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 16.7 [7.3 to 27.0] | 14.8 [7.9 to 25.8]

4. Secondary Outcome: Incidence of Skeletal Related Events
Description: Median time (in months) from randomisation until occurrence of a skeletal related event, where skeletal related event is defined as the first occurrence of a pathological fracture, a vertebral compression fracture not related to trauma, prophylactic surgery or radiation for impending fracture or spinal cord compression, or a spinal cord compression, using the Kaplan-Meier method.
Time Frame: From date of randomization until occurrence of a skeletal related event, assessed up to 31 months
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 18.4 [9.6 to 30.6] | 17.1 [9.3 to 25.8]

5. Secondary Outcome: Bone Metastases Formation
Description: Median time (in months) from randomisation to appearance of ≥4 new bone lesions using the Kaplan-Meier method
Time Frame: Patients were assessed every 12 weeks
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 15.1 [7.2 to 25.5] | 11.9 [7.0 to 22.5]

6. Secondary Outcome: Health Related Quality of Life
Description: Median time (in months) from randomisation until deterioration of Health related Quality of Life using the Kaplan-Meier method, where deterioration is defined as a change from baseline of less than or equal to -6 points in Total FACT-P score maintained for 2 consecutive visits.
Time Frame: Patients were assessed at every visit
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 5.5 [2.8 to 9.1] | 5.5 [2.8 to 9.1]

7. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Median time (in months) from randomisation to first PSA value >50% higher than baseline of at least 5ng/ml seen in at least 2 consecutive PSA values at least 2 weeks apart using the Kaplan-Meier method.
Time Frame: Patients were assessed every 12 weeks
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 5.6 [2.9 to 11.1] | 5.6 [2.8 to 11.4]

8. Secondary Outcome: Time to Pain Progression
Description: Median time (in months) from randomisation to first assessment of an increased pain event, where increased pain event is defined as the first of a patient requiring opiate medication for duration of ≥1 week for pain due to prostate cancer metastasis, pain due to metastasis that has an increase in the worst pain item of the Brief Pain Inventory (BPI) from baseline to a minimum score of 5 with no decrease in analgesic use, or pain due to metastasis requiring radionuclide therapy, radiation therapy or surgery.
Time Frame: Patients were assessed every 12 weeks
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 9.0 [3.3 to 19.4] | 8.4 [3.4 to 19.1]

9. Secondary Outcome: Time to Initiation of Chemotherapy
Description: Median time (in months) from randomisation to first administration of any chemotherapy using the Kaplan-Meier method
Time Frame: Patients were assessed every 12 weeks
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 299 | 295
Months | 11.4 [5.8 to 18.5] | 10.6 [6.0 to 18.2]

10. Secondary Outcome: Pharmacokinetic Characteristics of ZD4054
Time Frame: PK samples were performed at randomisation, Week 4, Week 8 and Week 12
Reporting Status: Not Posted
Measure: Least Squares Mean (95% Confidence Interval); unit: Plasma concentration versus time

ADVERSE EVENTS:
Arm/Group | ZD4054 | Placebo
Serious Adverse Events (participants affected / at risk) | 98/298 | 105/295
Other Adverse Events (participants affected / at risk) | 257/298 | 221/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 (N=298) | Placebo (N=295)
Anaemia (Blood and lymphatic system disorders) | 6 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 6 | 0
Myocardial Infarction (Cardiac disorders) | 3 | 2
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 1
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 1 | 1
Atrioventricular Block (Cardiac disorders) | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Prinzmetal Angina (Cardiac disorders) | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 2 | 7
Pyrexia (General disorders) | 3 | 2
Disease Progression (General disorders) | 1 | 2
Oedema Peripheral (General disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 1
Sepsis (Infections and infestations) | 3 | 3
Bronchopneumonia (Infections and infestations) | 2 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 2
Septic Shock (Infections and infestations) | 0 | 2
Abscess Jaw (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infected Cyst (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 1
Necrotising Fasciitis (Infections and infestations) | 1 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Post Procedural Infection (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Viral Pericarditis (Infections and infestations) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural Haematoma (Injury, poisoning and procedural complications) | 2 | 1
Cerebral Haemorrhage Traumatic (Injury, poisoning and procedural complications) | 0 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 1
Cystitis Radiation (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic Rupture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 3 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 2
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebral Thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular Disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss Of Consciousness (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 1 | 1
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1
Vith Nerve Paralysis (Nervous system disorders) | 0 | 1
Completed Suicide (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 4
Urinary Retention (Renal and urinary disorders) | 3 | 0
Renal Failure (Renal and urinary disorders) | 1 | 2
Anuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Haemorrhage Urinary Tract (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Urethral Stenosis (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 0 | 1
Prostatic Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 2
Aortic Dissection (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Iliac Artery Occlusion (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 (N=298) | Placebo (N=295)
Anaemia (Blood and lymphatic system disorders) | 46 | 33
Neutropenia (Blood and lymphatic system disorders) | 11 | 16
Nausea (Gastrointestinal disorders) | 62 | 44
Constipation (Gastrointestinal disorders) | 61 | 51
Diarrhoea (Gastrointestinal disorders) | 28 | 46
Vomiting (Gastrointestinal disorders) | 34 | 23
Oedema Peripheral (General disorders) | 132 | 56
Fatigue (General disorders) | 58 | 52
Pyrexia (General disorders) | 30 | 22
Asthenia (General disorders) | 18 | 22
Rhinitis (Infections and infestations) | 35 | 13
Nasopharyngitis (Infections and infestations) | 28 | 25
Urinary Tract Infection (Infections and infestations) | 19 | 24
Weight Decreased (Infections and infestations) | 15 | 13
Decreased Appetite (Metabolism and nutrition disorders) | 44 | 37
Back Pain (Musculoskeletal and connective tissue disorders) | 35 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 32
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 22 | 23
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 15 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 16
Headache (Nervous system disorders) | 92 | 37
Hypoaesthesia (Nervous system disorders) | 17 | 8
Dizziness (Nervous system disorders) | 14 | 16
Dysgeusia (Nervous system disorders) | 11 | 17
Insomnia (Psychiatric disorders) | 24 | 19
Haematuria (Renal and urinary disorders) | 20 | 19
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 48 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 19
Hypertension (Vascular disorders) | 11 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca can review results communications prior to public release and may within 60 days of receipt require amendments to be made. AstraZeneca can also require that submission or disclosure be delayed to allow for the filing of a patent application.